CLINICAL TRIAL: NCT00895609
Title: Dose Finding Study for Sugammadex and Neostigmine at Residual Neuromuscular Blockade (T4/T1 = 0.5)
Brief Title: Sugammadex and Neostigmine at Shallow Neuromuscular Blockade
Acronym: SUNDRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUNDRO
Record Dates: First submitted 2009-04-29; First posted 2009-05-08 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Neuromuscular Block
Keywords: Residual neuromuscular block; post-operative residual curarization; PORC; sugammadex; neostigmine; Shallow neuromuscular block (TOF-ratio of 0.5)
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugammadex (Experimental): Sugammadex in doses: 0 (placebo), 0.0625, 0.125, 0.25, 0.5 and 1 mg/kg
  Interventions: Drug: Sugammadex, Neostigmine, Saline
- Neostigmine (Active Comparator): Neostigmine in doses: 0 (placebo), 5, 8, 15, 25, 40 mg/kg
  Interventions: Drug: Sugammadex, Neostigmine, Saline

INTERVENTIONS:
Drug: Sugammadex, Neostigmine, Saline — Single intravenous injection of either:
  Sugammadex 0.0625 mg/kg (Sgx 0.0625) Sugammadex 0.125 mg/kg (Sgx 0.125) Sugammadex 0.25 mg/kg (Sgx 0.25) Sugammadex 0.5 mg/kg (Sgx 0.5) Sugammadex 1.0 mg/kg (Sgx 1.0) Neostigmine 5 mg/kg (Neo 5) Neostigmine 8 mg/kg (Neo 8) Neostigmine 15 mg/kg (Neo 15) Neostigmine 25 mg/kg (Neo 25) Neostigmine 40 mg/kg (Neo 40) Saline 0.9% (Saline)

SUMMARY:
This study is designed to compare recovery times after reversal of a residual neuromuscular block (TOF-ratio 0.5) with different doses of either neostigmine or sugammadex.

DETAILED DESCRIPTION:
Muscle relaxants are integral part of modern anesthesia. They optimize intubating conditions, reduce laryngeal trauma and improve operating conditions. Drawback is a possible pharmacological (muscle relaxing) effect of these drugs beyond the end of the operation (i.e. post-operative residual curarization: PORC). Reportedly about 30% of all patients who received muscle relaxants show signs of PORC when arriving in the post-anesthesia care unit. PORC comprises the risk of impaired post-operative fine motor and coordinative skills with a possible impairment of swallowing pharyngeal secretions with an increased risk of aspiration after extubation. Possible deleterious effects of this could be pneumonia, bronchitis, myocardial infarction, cardiac insufficiency, stroke or re-operation.

In order to avoid PORC patients with residual neuromuscular block receive a muscle relaxant antagonist from the anesthetist at the end of the operation. However, these drugs (neostigmine, pyridostigmine, etc.) from the class of cholinesterase inhibitors have unwanted effects such as bradycardia, increased gastro-intestinal motility, post-operative nausea and vomiting, salivation etc. To decrease these unwanted side effects cholinesterase inhibitors have to be given in combination with parasympatholyics e.g. atropine or glycopyrrolate with their own spectrum of unwanted side effects.

From October 2008 on, Sugammadex, a completely new reversal drug was introduced in to clinical practice. Sugammadex, is a modified gamma-cyclodextrine able to specifically bind rocuronium (a steroidal muscle relaxant). The complex is eliminated via the kidneys. However, all studies so far have focussed on reversal of profound or deep neuromuscular blockade. This study is designed to compare recovery times after reversal of a residual neuromuscular block (TOF-ratio 0.5) with different doses of either the neostigmine or sugammadex.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA physical status I - III
* Patients between 18 and 64 years
* Patients scheduled for general anesthesia with intubation using rocuronium
* Patients having given informed consent to the study

Exclusion Criteria:

* Anatomic and functional malformations with expected difficult intubation
* Known or suspected neuromuscular disease
* Significant hepatic or renal dysfunction
* Known or suspected history or family history of disposition to malignant hyperthermia
* Known or suspected allergy towards sugammadex, anesthetics, muscle relaxants, or other drugs used for general anesthesia
* Use of drugs that interfere with muscle relaxants
* Patients, included in another trial within the last 30 days
* Patients, with legal guidant
* Patients with contraindication towards the use of Sugammadex, neostigmine or glycopyrrolate
* Patients, which have already participated in a sugammadex trial
* Pregnant women (exclusion of pregnancy: postmenopausal status, negative β- HCG screen, status post tubal ligation)
* Breastfeeding women

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Time to TOF-ratio 0.9 following the investigational drug | Regular anesthesia time, approximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- [Background] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265